CLINICAL TRIAL: NCT06504602
Title: Pain Elimination and Anxiety Control Through Experiential Virtual Reality
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Los Angeles (Other)
Responsible Party: Principal Investigator, Matan Paret, Principal Investigator, Children's Hospital Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CHLA-24-00171
Record Dates: First submitted 2024-07-11; First posted 2024-07-17 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Procedural Pain; Procedural Anxiety
MeSH Terms: conditions — Pain, Procedural

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Active Virtual Reality (Experimental): Within the active virtual reality group virtual environment, participants will play the game Bearblast using Oculus Go Headset for patients 8-21 years old. In BearBlast, participants travel on a pre-set path through an interactive environment.
  Interventions: Device: Active Virtual Reality
- Passive Virtual Reality (Experimental): Within the passive virtual reality group virtual environment and age appropriate movie.
  Interventions: Device: Passive Virtual Reality
- Standard of Care (No Intervention): Participants will receive standard of care distraction methods.

INTERVENTIONS:
Device: Active Virtual Reality — Active virtual reality group will play a game through a virtual environment.
  Arms: Active Virtual Reality
Device: Passive Virtual Reality — Passive virtual reality group will watch a movie through a virtual environment.
  Arms: Passive Virtual Reality

SUMMARY:
The goal of this clinical trial is to determine if active virtual reality is more effective than passive virtual reality and standard of care distraction in decreasing pain in children, from 8 to 21 years old, undergoing intravenous placement in emergency department. The main question[s] it aims to answer [is/are]:

* Will active virtual reality reduce pain score on Faces Pain Scale - revised and measure of heart rate during intravenous placement for children ages 8 years old to 21 years old more than passive virtual reality and standard of care?
* Will active virtual reality reduce anxiety score on Visual Analog Scale - revised and measure of heart rate during intravenous placement for children ages 8 years old to 21 years old more than passive virtual reality and standard of care?

If there is a comparison group: Researchers will compare active group to passive group and standard of care.

Participants will randomized into active virtual reality, passive virtual reality or standard of care arms.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents 8-21 years old undergoing IV placement .

  * Ability to understand study procedures and to comply with them for the entire length of the study.
  * Participants and caregiver speaking English or Spanish.

Exclusion Criteria:

* Participants with psychiatric, developmental delay, visual or auditory deficits that would interfere with virtual reality gameplay (decision based on treating clinicians' evaluation).

  * Participants receiving narcotics, opioids, or anxiolytics 8 hours prior (Tylenol and ibuprofen do not count).
  * Participants with pain so significant that consent/assent is not possible (decision based on treating clinician evaluation).
  * Critically ill Participants (ESI 1).

Ages: 8 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 96 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-03-15 (Estimated); Study Completion 2025-03-15 (Estimated)

PRIMARY OUTCOMES:
Mean Change from Baseline in Pain Scores on Faces Pain Scale - Revised after IV Placement | 5 minutes before, immediately after procedure
  Pain score on Faces Pain Scale - Revised will be assessed 5 minutes before and immediately after procedure. The minimum score is 0, and the maximum score is 10. Higher scores correlate to a worse outcome (more pain).

SECONDARY OUTCOMES:
Mean Change from Baseline in Anxiety Scores on Visual Analog Scale after IV Placement | 5 minutes before, immediately after procedure
  Anxiety score on Visual Analog Scale will be assessed 5 minutes before and immediately after procedure. The minimum score is 0, and the maximum score is 100. Higher scores correlate to a worse outcome (more anxiety).
Mean Change from Baseline in Heart Rate after IV Placement | 5 minutes before, during, and immediately after procedure
  Heart Rate will be measured 5 minutes before, during, and immediately after procedure

CONTACTS AND LOCATIONS:
Overall Officials: Matan Paret, MD, Principal Investigator — Children's Hospital Los Angeles

IPD SHARING:
Plan to Share IPD: No